CLINICAL TRIAL: NCT05402839
Title: Molecular Genetics Study on Screening of Malignant Hyperthermia Susceptible Individuals
Brief Title: Screening of Malignant Hyperthermia Susceptible Individuals
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Guo Xiangyang, Chief of the department of anesthesiology, Peking University Third Hospital
Other Study IDs: MR-11-22-002000
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Malignant Hyperthermia
MeSH Terms: conditions — Malignant Hyperthermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study intends to target patients who underwent surgery under general anesthesia during the study period and developed malignant hyperthermia during or after surgery. Therefore, the total sample size was estimated to be about 50 people based on the past incidence of this rare disease. Every year, about 20 patients and their families who developed malignant hyperthermia during or after surgery will participate in this nationwide study (estimated by the current incidence of malignant hyperthermia), and about 1-5 patients will be admitted to Peking University Third Hospital participate in this research. Relevant specimens were collected from malignant hyperthermia (MH) patients and their family members for genetic analysis to determine the mutation of MH-related pathogenic gene loci.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery under general anesthesia during the study period developed malignant hyperthermia during or after surgery.

Exclusion Criteria:

* Malignant hyperthermia was ruled out by later treatment and diagnosis;
* The patient or family member refuses to be recruited.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Since the incidence of malignant hyperthermia is low (1/50,000 in adults, 1/15,000 in children), it is a rare disease, so this study will continue for 10-20 years. This study is an observational study, so the sample is estimated based on the past incidence of this rare disease. The amount is about 50 patients.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2041-02 (Estimated); Study Completion 2041-02 (Estimated)

PRIMARY OUTCOMES:
Whole exome sequencing | immediately after MH was diagnosed

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China